CLINICAL TRIAL: NCT06852794
Title: USE OF ARTIFICIAL INTELLIGENCE IN THE BACK-OFFICE OF A SPECIALIZED MEDICAL CLINIC FOR PULMONARY FIBROSIS (LLM-ILD)
Brief Title: USE OF ARTIFICIAL INTELLIGENCE IN A PULMONARY FIBROSIS CLINIC
Acronym: LLM-ILD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7002
Record Dates: First submitted 2025-01-30; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Disease
Keywords: Artificial Intelligence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients attending ILD clinic (Experimental)
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The patients will receive questionnaires. The enrolled patients will be asked to provide feedback on the answers they read.

SUMMARY:
The present study aims to evaluate the usefulness of artificial intelligence (AI) in the back-office of an ILD (Interstitial Lung Disease) clinic.

ELIGIBILITY:
Inclusion Criteria:

- Patients attending ILD clinic of the IRCCS Fondazione Policlinico A. Gemelli.

Exclusion Criteria:

* Patients unable or unwilling to sign the informed consent
* Patients who are senders of one of the emails chosen for the questionnaire
* Patients with manifest inability to fill out the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Variation of VAS scores of clarity of the message in questionnaires administered at T1 and at T2 | 15 days
Variation of VAS scores of empathy conveyed in questionnaires administered at T1 and at T2 | 15 days

SECONDARY OUTCOMES:
Percentage of answers recognised correctly as answers provided by AI among the total of answers flagged as provided by AI by study subjects | 1 day
Stratify the results by patients' demographic characteristics and past experiences with artificial intelligence systems. | 1 day